CLINICAL TRIAL: NCT07168369
Title: The Effect of Early Nutritional Intervention on Muscle Mass in Patients Who Have Undergone Liver Transplantation
Brief Title: Early Nutritional Intervention in Patients Undergoing Liver Transplantation
Acronym: NutLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-238; 21-371
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2020-10

CONDITIONS: Liver Transplant
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received a protein and energy-rich supplement (1 bottle of 235mL per day for 12 weeks) in addition to standard care.
  Interventions: Dietary Supplement: protein and energy-rich supplement
- Control group (No Intervention): The control group received standard care, which consists of a meeting with a registered dietitian providing routine dietary advice after surgery.

INTERVENTIONS:
Dietary Supplement: protein and energy-rich supplement — The nutritional supplements were provided in the form of ready-to-drink liquid solutions rich in protein and energy. Patients without diabetes received one 235 ml bottle per day of Ensure® Protéine Max (Abbott Nutrition, Montreal, Canada), which contained 350 kcal, 20 g of protein, 11 g of fat, 44 g of carbohydrates, 1.5 g of calcium-HMB and other essential micronutrients. Patients diagnosed with diabetes prior to LT received one 237 ml bottle per day of Boost® Diabetic (Nestlé, Montreal, Canada), which provided 190 kcal, 16 g of protein, 7 g of fat, 17 g of carbohydrates, and other essential micronutrients. Patients were instructed to consume the supplement in four equal doses of ~60 ml each, taken daily with breakfast, lunch, dinner, and as a bedtime snack, totaling one full bottle per day. The supplementation lasted for 12 weeks, beginning once solid oral feeding was initiated.
  Arms: Intervention group

SUMMARY:
The main goal of this clinical study is to assess the feasibility of a 12-week oral nutritional supplementation post-liver transplantation (LT). Secondary objectives includes evaluating changes in nutritional risk, muscle strength and mass, and quality of life during the pre-transplant period, as well as the intervention's potential impact post-LT. Following LT, participants are randomized to either: a control group, or an intervention group (high protein and energy oral supplement (235mL) for 12 week). Participants awaiting LT will complete questionnaires including nutritional risk (Liver Disease Undernutrition Screening Tool), muscle strength (Chair Stand Test), and quality of life (SF-36) every three months until surgery, at discharge after LT, and at 12 weeks. Muscle mass is measured by a computed tomography (CT) scan at admission for LT and at 12 weeks. Feasibility is assessed via eligibility rate, recruitment rate, target recruitment rate, protocol and intervention adherence, attrition rate, and safety.

ELIGIBILITY:
Inclusion Criteria:

* patients with cirrhosis listed for LT
* French or English speaking

Exclusion Criteria:

* patients awaiting multiple organ transplants
* patients with acute liver failure or hepatocellular carcinoma
* patients who stayed in the intensive care unit for more than 30 days after LT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Study feasibility | From enrollment to the end of treatment at 12 weeks
  Feasibility of the study was assessed using a set of predefined indicators: the eligibility rate (% of patients on the waiting list who met eligibility criteria), the recruitment rate (% of eligible patients who agreed to participate), the target recruitment rate (% of participants enrolled relative to the predefined sample size), adherence to the protocol (% of participants who completed all planned data collection time points), and adherence to the intervention (% of participants who followed the nutritional intervention as intended). The attrition rate was also measured as the percentage of participants lost to follow-up or withdrawn after LT. The incidence of serious and non-serious adverse events during the study period was documented to evaluate the safety of the intervention.

SECONDARY OUTCOMES:
Nutritional risk | From enrollment to the end of treatment at 12 weeks
  The nutritional risk of participants was assessed using the Liver Disease Undernutrition Screening Tool (LDUST), which is specifically designed for patients with chronic liver disease. This tool includes six questions addressing nutritional intake, weight loss, subcutaneous fat loss, muscle mass loss, fluid accumulation, and reduced functional capacity. The LDUST has shown good correlation with dietitian assessments of malnutrition. Using the LDUST, patients were classified into one of two categories: absence or presence of malnutrition risk.
Muscle strength | From enrollment to the end of treatment at 12 weeks
  Muscle strength was assessed using the Chair Stand Test (CST), which provides a functional evaluation of muscle strength and endurance. The CST allows for a robust measure of lower limb function. Starting from a seated position, participants were asked to stand up and sit down without using their arms (the participant's arms were crossed over their chest) for a total of five times without assistance. The test was performed three times, and the average completion time was recorded. Patients unable to perform the test were assigned a score of 32 seconds. A completion time exceeding 15 seconds indicates reduced muscle strength
Muscle mass | At admission for LT and at the end of treatment at 12 weeks
  Muscle mass was assessed using SMI measured by CT scan, the gold standard method for quantitative evaluation of sarcopenia. The skeletal muscle area was measured in cm2 from CT by segmenting muscles at the level of the third lumbar vertebra (L3) and normalized to height in m2. The SMI at the L3 level has demonstrated a strong correlation with clinical outcomes and with total body muscle mass. A SMI of less than 38.5 cm²/m² for women and less than 52.4 cm²/m² for men were used as cut-off values to define reduced muscle mass in this study. As recommended by EWGSOP, the diagnosis of sarcopenia was based on low SMI combined with reduced muscle strength, assessed using the CST.
Health-related quality of life | From enrollment to the end of treatment at 12 weeks
  Quality of life was assessed using the Short Form 36 (SF-36) questionnaire, a validated and widely used tool for evaluating participants' perceptions of their quality of life. The SF-36 consists of 36 questions and covers 8 health dimensions: physical activity, limitations due to physical condition, limitations due to mental health, life and social relations, pain, vitality, mental health, and perceived health. Responses are scored from 0 to 100, with each dimension comprising 2 to 10 questions. The domain scores are further grouped into overall physical and mental health scores. Additionally, the SF-36 includes a question related to the evolution of health perceived by the patient. Higher scores reflect better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche du Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No